CLINICAL TRIAL: NCT03056196
Title: Age-Adjusted D-Dimer and Two-Site Compression POINt-OF-CARE Ultrasonography to Rule Out Acute Deep Vein Thrombosis
Brief Title: Two-Site Compression POINt-OF-CARE Ultrasonography for DVT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Khalifa Alqaydi, senior resident in emergency medicine, Jewish General Hospital
Other Study IDs: 17-010
Record Dates: First submitted 2017-02-09; First posted 2017-02-17 (Actual); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Deep Vein Thrombosis; Point of Care Ultrasound
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: point of care ultrasound — want to assess the ability of d-dimer test and point of care ultrasound to role out lower leg DVT

SUMMARY:
Introduction

Undiagnosed deep vein thrombosis (DVT) can lead to significant morbidity and mortality, including death from DVT-associated massive pulmonary embolism (PE). While several validated clinical prediction rules, blood test and imaging modalities exist to investigate a potential DVT, there is currently a lack of rapid, accessible and reliable methods to exclude the possibility of DVT without resorting to formal venous duplex scanning.

Currently, the use in the ED of a validated clinical prediction rule combined with high-sensitivity D-dimer test has a poor predictive value, as 75-90% of patients suspected of DVT have a negative formal venous duplex scan.

Compression bedside ultrasound has however recently been shown to be a safe, rapid and accurate method for the diagnosis of proximal DVT in the emergency department with a high sensitivity and specificity (combined sensitivity and specificity of 96.1% and 96.8%, respectively1).

Research Question

In the present study, the investigators will primarily assess whether two-site compression POCUS combined with a negative age-adjusted D-dimer test can accurately rule out DVT in ED patients regardless of the Wells criteria.

Methods

This is a single-center, prospective, observational study carried out over one year in the Emergency Department of the Jewish General Hospital in Montreal, Quebec. The investigators aim to enroll a convenience sample of 475 patients aged 18 years and older presenting to the ED with symptoms suggestive of a DVT. All enrolled patients will receive the standard of care required for a lower leg DVT presentation. After calculating Patients DVT risk using modified wells criteria, all patients will undergo POCUS for DVT followed by a D-dimer test. Based on their results, patients will either undergo formal duplex scanning, or will be discharged without further testing and receive a three-month phone follow-up.

A true negative lower leg DVT will be defined as follows:

1. Negative follow-up phone questionnaire for patients who were sent home with no formal duplex venous scanning.
2. Negative formal duplex venous scanning for patients who were deemed likely to have lower leg DVT using the Wells score, with a negative D-dimer and POCUS

Age-adjusted DVT was added to account for below knee DVT and avoid the need for patients to return for fellow up duplex study in 1 week.

To estimate our technique's sensitivity with a 4% margin of error with 95% confidence intervals, 92 confirmed DVT patients are needed. The investigators expect to recruit a total 475 patients within one-year period at the JGH (95 DVT-positive patients and 380 DVT-negative patients).

Impact

The use of compression bedside ultrasound with a negative age-adjusted D-dimer test to rule out DVT in the ED may accelerate the decision regarding patient disposition and significantly decrease the length of patient stay in the ED. In addition, it may help avoid unnecessary medical interventions and diagnostic tests, thus representing potential quality of care and cost-saving improvements as well.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 years and older presenting to the ED with symptoms suggestive of a DVT

Exclusion Criteria:

* Pregnancy
* Recent traumatic injury to the lower extremity
* Hemodynamic instability
* Suspected pulmonary embolism
* CT angiography (pulmonary embolism protocol including lower extremities) performed before ED POCUS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients aged 18 years and older presenting to the ED with symptoms suggestive of a DVT
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-03-01 (Estimated); Primary Completion 2018-02-28 (Estimated); Study Completion 2018-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants who can have the diagnosis of DVT excluded using two-site compression POCUS combined with a negative age-adjusted D-dimer regardless of the Wells criteria. | 1 year

IPD SHARING:
Plan to Share IPD: No
Not going to share patients data